CLINICAL TRIAL: NCT06109220
Title: Clinical Study on the Safety and Efficacy of Intrarticular Injection of Autologous Adipose-derived Vascular Matrix Components (SVF) in the Treatment of Knee Osteoarthritis (KOA)
Brief Title: Treatment of Knee Osteoarthritis (KOA) by Injection of Autologous Adipose-derived Vascular Matrix Components (SVF) Into Joint Cavity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KY20232112-X-1
Record Dates: First submitted 2023-08-18; First posted 2023-10-31 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-03

CONDITIONS: Knee Osteoarthritis
Keywords: Stromal vascular fraction
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Stage of arthritis (Experimental): Patients with unilateral or bilateral knee degenerative inflammation (KOA) with Kellgren-lawrence rating of level 3 or lower
  Interventions: Behavioral: Stromal vascular fraction,SVF

INTERVENTIONS:
Behavioral: Stromal vascular fraction,SVF — SVF was injected into the knee cavity

SUMMARY:
The purpose of this study was to analyze and study the efficacy and safety of autologous adipose-derived vascular matrix components (SVF) in patients with knee osteoarthritis before and after treatment through clinical evaluation, radiation index, and metabolic index comparison between plasma and irrigation solution before and after SVF injection.

ELIGIBILITY:
Inclusion Criteria:

* The age range is 20-70 years old
* Patients with unilateral or bilateral knee degenerative inflammation (KOA) with Kellgren-lawrence rating of level 3 or lower
* The physical health status is mainly in the ASA grade Ⅰ, Ⅱ and Ⅲ
* Subjects had no active tumors, no active inflammation, no treponema pallidum, HIV, hepatitis B virus, or hepatitis C virus
* The subject shall provide the physical examination report of knee X-ray examination, MRI examination and other items

Exclusion Criteria:

* Patients with nonunion or displaced fractures around defective cartilage
* Pregnant or lactating women
* Autoimmune disease
* Subjects with diabetes (exceptions are patients whose blood sugar levels remain within the normal range and diabetes has not caused other complications)
* The patients had severe neurological diseases affecting the evaluation of postoperative results

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-03-30 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
T2 mapping | 24 months after the first SVF injection into the knee cavity
  The degree of change of articular cartilage was observed

SECONDARY OUTCOMES:
Western Ontario and McMaster Universities Arthritis Index (WOMAC) | 24 months after the first SVF injection into the knee cavity
  The WOMAC is a specific assessment scale for osteoarthritis, which is assessed according to three aspects: pain, stiffness and function. A total of 24 WOMAC scores were scored, 0-10 points for each item, with a total score of 240 points. A total score <80 was mild OA, a total score of 80-120 was moderate OA, and a total score of >120 was severe OA.The severity and therapeutic effect of arthritis were evaluated according to the relevant symptoms and signs of patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Xijing Hospital, Xi'an, Shannxi, China

IPD SHARING:
Plan to Share IPD: No